CLINICAL TRIAL: NCT06131892
Title: Defibrillation in Accidental Hypothermia: a Retrospective Study of the International Hypothermia Registry
Brief Title: Defibrillation in Accidental Hypothermia
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Evelien Cools, Medical Doctor, Principal Investigator, University Hospital, Geneva
Other Study IDs: 2023-01087
Record Dates: First submitted 2023-10-22; First posted 2023-11-14 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Hypothermia, Accidental; Defibrillation
MeSH Terms: conditions — Hypothermia | interventions — Electric Countershock

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Successful defibrillation during extra corporeal life support (ECLS) rewarming
  Interventions: Other: Defibrillation
- Non Successful defibrillation during extra corporeal life support (ECLS) rewarming
  Interventions: Other: Defibrillation
- Successful defibrillation before rewarming or during non-ECLS rewarming: non- ECLS: non- extra corporeal life support
  Interventions: Other: Defibrillation
- Non- successful defibrillation before rewarming or during non-ECLS rewarming: non- ECLS: non- extra corporeal life support
  Interventions: Other: Defibrillation

INTERVENTIONS:
Other: Defibrillation — Defibrillation

SUMMARY:
Hypothermia (core temperature ≤35°C) is a frequent and life-threatening complication after mountain accidents, near-drowning, and intoxications, and can provoke arrhythmia, reduced cardiac contractility, and cardiac arrest. The hypothermic heart may be insensitive to defibrillation with a core temperature <30°C. Also, below <30°C after successful defibrillation, a perfusing rhythm often degenerates to ventricular fibrillation (VF) again. Repeated defibrillation can induce myocardial injury. Thus, the guidelines of the European Resuscitation Council (ERC) suggest delaying further defibrillation attempts until the core temperature is >30°C if VF persists after 3 shocks. Epinephrine should be withheld if core temperature is <30°C. Advanced Life Support (ALS) guidelines of the American Heart Association (AHA) state that it may be reasonable to perform further defibrillation attempts according to the standard algorithm and to consider administration of a vasopressor during cardiac arrest (Table 1). This discrepancy between ERC and AHA guidelines can be explained by the different interpretations of mainly animal data, which show that vasopressors increase the chances of successful defibrillation <30°C, defined as return of spontaneous circulation (ROSC) for at least 30 seconds. The guidelines of the Wilderness and Environmental Medicine Society (WMS) state that a single shock at a maximum power can be given for patients with a temperature <30°C.

The aim of this study is to evaluate clinical course of hypothermic patients(<30°C) undergoing defibrillation. The primary aim is to evaluate the success ratio of defibrillation, defined as ROSC for at least 30 seconds. Secondary aims are the recurrence rate of ventricular fibrillation, the number of defibrillation attempts per patient, the presence of cardiac dysfunction after defibrillation and the cerebral performance category (CPC) score at the end of hospitalization.

ELIGIBILITY:
Inclusion Criteria:

- patients of the International Hypothermia Registry with a defibrillation while having a body core temperature equal or less than 30°C

Exclusion Criteria:

* patients of the International Hypothermia Registry with a body core temperature >30°C
* patients who refused to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with accidental hypothermia and a body core temperature equal or less than 30°C who had one or more defibrillation attempts
Sampling Method: Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
the number of patients with a core temperature equal or less than 30°C who had a successful defibrillation, defined as ROSC for at least 30 seconds | through study completion, an average of 3 months

SECONDARY OUTCOMES:
the number of patients with a return to ventricular fibrillation after successful defibrillation | through study completion, an average of 3 months
the rate of defibrillation attempts per patient | through study completion, an average of 3 months
the number of patients with the presence of cardiac dysfunction after defibrillation | through study completion, an average of 3 months
  a decrease in cardiac output, or a reduced ejection fraction, systolic or diastolic dysfunction on echocardiographic ultrasound
cerebral performance category (CPC) score of every patient at the end of hospitalization | through study completion, an average of 3 months
  a score from 1 to 5, with "1" meaning "Good Outcome", "5" means dead

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Anaesthesiology, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No